CLINICAL TRIAL: NCT00233766
Title: An Evaluation of Two Reduced Sirolimus Doses on the BX VELOCITY Balloon-Expandable Stent in the Treatment of Patients With de Novo Native Coronary Artery Lesions(REDOX)
Brief Title: Evaluation of Two Reduced Sirolimus Doses in Treatment of de Novo Coronary Artery Lesions (REDOX)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: J. E. Sousa, MD, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02-6314
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Bx VELOCITY Stent containing 45% and 70% of Sirolimus dose

SUMMARY:
The objective of this study is to assess the performance and safety of two reduced sirolimus doses on the Bx VELOCITY Balloon-Expandable stent, mounted on the Raptorâ rapid exchange (RX) Stent Delivery System (SDS) in patients with de novo native coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female patient minimum 18 years of age
2. No significant (>50%) untreated stenoses proximal or distal to the target lesion that will not be treated during the procedure and may require revascularization or impede runoff;
3. Target lesion is 18mm in length (visual estimate);
4. Target lesion is 3.0mm and 3.5mm in diameter (visual estimate);
5. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. A Q-wave or non-Q-wave myocardial infarction within the preceding 72 hours unless the CK and CK-MB enzymes are back to normal;
2. Ejection fraction 30%;
3. Stent placement of target lesion covers a side branch >2.0mm in diameter;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Late loss measured by quantitative coronary angiography at four-months and twelve-months post-procedure. | four-months and twelve-months post-procedure
NIH volume as measured by intravascular ultrasound (IVUS) at four-months and twelve-months post-procedure. | four-months and twelve-months post-procedure
Volumetric plaque burden as measured by IVUS at four-months and twelve months post-procedure. | four-months and twelve months post-procedure
Four and twelve month target vessel failure (TVF). | Four and twelve month

CONTACTS AND LOCATIONS:
Overall Officials: J. E. Sousa, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil

REFERENCES:
- [Background] Nakamura M, Abizaid A, Hirohata A, Honda Y, Sousa JE, Fitzgerald PJ. Efficacy of reduced-dose sirolimus-eluting stents in the human coronary artery: serial IVUS analysis of neointimal hyperplasia and luminal dimension. Catheter Cardiovasc Interv. 2007 Dec 1;70(7):946-51. doi: 10.1002/ccd.21272. PMID 17621671